CLINICAL TRIAL: NCT03693066
Title: Effectiveness of the Ozone Application in Two-Visit Indirect Pulp Therapy of Permanent Molars With Deep Carious Lesion
Acronym: ozone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Merve AKCAY, assoc prof dr, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 213S004
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Ozone; Caries
Keywords: stepwise excavation; indirect pulp capping; ozone; deep caries
MeSH Terms: interventions — Ozone; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ozone (Experimental): Thirty five molar teeth with deep caries lesion were selected to apply two-visit indirect pulp therapy with ozone. The peripheral demineralized dentin and the superficial necrotic dentin were completely removed, and left some caries at the central part. The cavity was exposed to gaseous ozone for 60 seconds, with an ozone delivery system. The remaining caries dentin was covered with calcium hydroxide base material and cavity sealed with glass ionomer cement to reopen 4 months later.
  Interventions: Other: Ozone
- chlorhexidine digluconate (Active Comparator): Thirty five molar teeth with deep caries lesion were selected to apply two-visit indirect pulp therapy with chlorhexidine digluconate. The peripheral demineralized dentin and the superficial necrotic dentin were completely removed, and left some caries at the central part. Following the excavation, 2% chlorhexidine digluconate was applied to the cavity for 60 seconds using a brush. According to the manufacturer instructions, puddled solution was removed with a new brush without dry to leave site moist. The remaining caries dentin was covered with calcium hydroxide base material and cavity sealed with glass ionomer cement.
  Interventions: Other: chlorhexidine digluconate
- Control (Active Comparator): Thirty five molar teeth with deep caries lesion were selected to apply conventional two-visit indirect pulp therapy (control). The peripheral demineralized dentin and the superficial necrotic dentin were completely removed, and left some caries at the central part. The remaining caries dentin was covered with calcium hydroxide base material and cavity sealed with glass ionomer cement.
  Interventions: Other: Control

INTERVENTIONS:
Other: Ozone — In the two-visit indirect pulp therapy, due to reduce the number of bacteria remaining in the cavity, the antimicrobial agents can be used as cavity disinfectants such as ozone.
  Arms: ozone
Other: chlorhexidine digluconate — In the two-visit indirect pulp therapy, due to reduce the number of bacteria remaining in the cavity, the antimicrobial agents can be used as cavity disinfectants such as chlorhexidine digluconate.
  Arms: chlorhexidine digluconate
Other: Control
  Other Names: without any cavity disinfectant
  Arms: Control

SUMMARY:
The aim of this study was to evaluate the clinical and microbiological effectiveness of the ozone application in two-visit indirect pulp therapy.

Materials and Methods: One hundred and five lower first molar teeth with deep caries lesion were included and randomly assigned three groups to apply two-visit indirect pulp therapy. Treatment procedure was applied without any disinfectant(control), with 60s 2% chlorhexidine digluconate(CHX) or 60s ozone application. In four different stage (after initial excavation, ozone/CHX application before the temporary restoration, four months later immediately after removing temporary restoration, and final excavation) dentin humidity, consistency and colour properties were recorded to evaluate the clinical characteristics of the tissue, and standard dentin samples were collected for the microbiological analysis of mutans streptococci, lactobacilli and the total number of colony forming units. The data were analyzed by using Mann-Whitney-U test for multiple comparisons.

DETAILED DESCRIPTION:
A randomized, controlled, clinical trial was designed to evaluate the antibacterial effect of ozone application in two-visit indirect pulp therapy. The sample size for this study was determined 35 for each group (%82 power, 0.50 significance level). This study conducted with 49 female and 56 male patients aged between 6-13 years old (average 9.72). The entire patient had deep caries lesions with pulp perforation risk at one of the lower first permanent molars.

The vitality of teeth were tested by cold thermal test, necessary clinical and radiographic examinations were performed, then the teeth were randomly divided into three treatment groups as: two-visit indirect pulp therapy without any disinfectant (control group), two-visit indirect pulp therapy with chlorhexidine digluconate application (positive control group), and two-visit indirect pulp therapy with gaseous ozone application (experimental group). Treatment procedure started with the local anesthesia and isolation of the tooth with rubber-dam. The peripheral demineralized dentin and the superficial necrotic dentin were then completely removed, and left some caries at the central part. It was decided to leave potentially remineralizable affected dentin by hand sensitivity. In control group, the remaining caries dentin was covered with calcium hydroxide base material and cavity sealed with glass ionomer cement temporarily. In positive control group, following the excavation, 2% chlorhexidine digluconate was applied to the cavity for 60 seconds using a brush. According to the manufacturer instructions, puddled solution was removed with a new brush without dry to leave site moist. In experimental group, following the excavation, the cavity was exposed to gaseous ozone for 60 seconds, with an ozone delivery system. According the manufacturers, HealOzone produces ozone at a fixed concentration of 2,100 ppm. Ozone production is stopped if the airtight seal over the tooth is broken during treatment, therefore, silicon caps were selected according to the size of each tooth. After the disinfectant applications, procedure was completed as aforementioned in the control group for these two groups. After four months, the clinical and radiographic examinations were repeated in order to assess pathological conditions of the teeth before removed the temporary glass ionomer cement and calcium hydroxide base material. Subsequent to this procedure, remaining demineralized dentin was completely removed in all groups. Floor of the cavity was then covered with calcium hydroxide base material and glass ionomer cement as liner. Final restorations were performed with 2-stage self etch bond and composite.

For the clinical analyses, the consistency, colour and humidity of the dentine were recorded at three times: after initial excavation at the first stage (T0), at the end of four months period, immediately after removing the calcium hydroxide base at second stage (T2) and after final excavation at second stage (T3). The consistency of dentin was determined by probing and classified as; very soft, soft, medium hard and hard [8]. The colour of dentin was classified as, light yellow, yellow, light brown, dark brown/black. In addition, dentine was probed and if moisture leakage was occurred, it was classified as wet or if did not it would be classified as dry.

For the microbiological analyses, dentine samples were taken at four different times: from the remain dentine after initial excavation (T0), immediately after ozone/chlorhexidine application (T1), at the end of four months period immediately after removing the calcium hydroxide base material (T2) and after final excavation (T3). T1 stage did not exist in control group, because in this group no disinfectant was used. Clinical photographs were taken to ensure that all samples were collected from the same site in all following stages. The dentine samples were collected enough to fill the slots of a sterile No.16 round carbide bur (SS White Burs, Inc., New Jersey, USA) and the samples were placed into 1 ml thioglucolate medium and transported the microbiology laboratory in 2 hours to be analyzed for the mutans streptococci, lactobacilli and the total number of colony forming units (CFU).

The samples were homogenized on a vortex mixer for 15 seconds under laboratory conditions. Mitis Salivarius agar as the selective medium for Streptoccus mutans, Rogossa agar for Lactobacilli and Brain Hearth agar supplemented %5 blood for the total numbers of CFU were used. Samples were incubated anaerobically for 48 hours and the colonies were counted.

ELIGIBILITY:
Inclusion Criteria:

* Without signs of irreversible pulpitis (spontaneous pain, prolonged pain response etc.)
* The absence of percussion or palpation sensitivity, pathological mobility, or infection symptoms like fistula or abscess or discoloration in the clinical examination;
* Presence of normal lamina dura and periodontal range, absence of lesion, internal or external resorption or calcification in or around the root in the radiological examination.

Exclusion Criteria:

* Children with special health care needs
* Children with dental crowding limiting the child's ability to maintain oral hygiene
* Teeth with clinical and/ or radiological signs or symptoms of non- vitality
* Teeth with clinical and radiological signs or symptoms of irreversible pulpitis, or dental abscess (Pain, mobility, tenderness to percussion, draining sinus, pulp polyp, furcal or periapical radiolucency, root resorption)

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Changes microbiological count: from baseline to 4 months | Baseline and Four months later
  mutans streptococci, lactobacilli and the total number of colony forming units were counted.

SECONDARY OUTCOMES:
Changes characteristics of the dentin humidity: from baseline to 4 months | Baseline and Four months later
  Dentine was probed and if moisture leakage was occurred, it was classified as wet or if did not it would be classified as dry.
Changes characteristics of the dentin consistency: from baseline to 4 months | Baseline and Four months later
  The consistency of dentin was determined by probing and classified as; very soft, soft, medium hard and hard.
Changes characteristics of the dentin color: from baseline to 4 months | Baseline and Four months later
  The colour of dentin was classified as, light yellow, yellow, light brown, dark brown/black.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Akcay, assoc prof, Principal Investigator — Izmir Katip Celebi Uni

IPD SHARING:
Plan to Share IPD: Undecided